CLINICAL TRIAL: NCT07262957
Title: Preventing Postoperative Complications in Patients Undergoing High-risk Pancreatoduodenectomy With a Bundle Approach Including Hydrocortisone, Octreotide, and the Teres Ligament Patch (PANENCA): an International Randomized Controlled Multicenter Trial
Brief Title: Preventing Postoperative Complications in Patients Undergoing High-risk Pancreatoduodenectomy With a Bundle Approach Including Hydrocortisone, Octreotide, and the Teres Ligament Patch (PANENCA)
Acronym: PANENCA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Erasmus Medical Center (Other); UMC Utrecht (Other); Medisch Spectrum Twente (Other); Jeroen Bosch Ziekenhuis (Other); Maastricht University Medical Center (Other); Radboud University Medical Center (Other); Isala (Other); Catharina Ziekenhuis Eindhoven (Other); Helsinki University Central Hospital (Other); Oslo University Hospital (Other); Karolinska University Hospital (Other); Sahlgrenska University Hospital (Other); University Hospital, Linkoeping (Other); Lund University Hospital (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); Azienda Ospedaliera di Padova (Other); San Raffaele University Hospital, Italy (Other); Leiden University Medical Center (Other); University Medical Center Groningen (Other); Clinical Cancer Hospital, Kyiv (Other); Rigshospitalet, Denmark (Other); University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, M.G. Besselink, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-519667-18-00
Record Dates: First submitted 2025-11-25; First posted 2025-12-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pancreas Head Cancer; Pancreas Adenocarcinoma; IPMN, Pancreatic; Cholangio Carcinoma; Ampulla of Vater Adenocarcinoma; PDAC - Pancreatic Ductal Adenocarcinoma; Duodenal Carcinoma; Mucinous Cystic Neoplasm; Neuro Endocrine Tumours; Pancreatitis
Keywords: Whipple; Pancreatoduodenectomy; POPF; Major complications; Fistula; ISGPS; Hydrocortisone; Octreotide; Ligament teres patch
MeSH Terms: conditions — Pancreatic Intraductal Neoplasms; Duodenal Neoplasms; Pancreatitis; Fistula | interventions — Hydrocortisone; Octreotide

STUDY DESIGN:
Intervention Model Description: The PANENCA trial is an international, multicenter, randomized controlled trial with 1:1 parallel allocation to the intervention group (HOP bundle) or the control group (standard care).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (HOP bundle) (Experimental): Patients in the intervention group will receive the HOP bundle approach:
  a combination intervention of: Hydrocortisone, octreotide and the ligamentum teres patch
  Interventions: Combination Product: HOP bundle
- Controle arm (No Intervention): Standard care

INTERVENTIONS:
Combination Product: HOP bundle — Patients in the intervention group will receive the HOP bundle approach:
  * Hydrocortisone intravenous: 100mg hydrocortisone as sodium succinate i.v. starting during the induction of general anesthesia, administered every 8 hours until 2 days perioperative (last dose evening postoperative day 2) (total 9 dosages).
  * Octreotide subcutaneous: 0,1 mg every 8 hours during maximum 7 days, starting during the induction of general anesthesia, administered minimal 1 hour before surgery (to a maximum of 21 dosages or until earlier discharge).
  * Intraoperative coverage of the gastroduodenal artery stump using a teres ligament patch, separating it from the pancreato-enteric anastomosis.
  Other Names: Hydrocortisone; Octreotide; Ligament teres patch
  Arms: Intervention arm (HOP bundle)

SUMMARY:
The PANENCA trial aims to reduce postoperative complications in patients undergoing pancreatoduodenectomy (also known as a Whipple procedure), a complex surgical operation performed to remove tumors located in or near the head of the pancreas. One of the most frequent and serious complications after this surgery is postoperative pancreatic fistula (POPF), a leakage of pancreatic fluid from the surgical connection. POPF can lead to intra-abdominal infection, bleeding, and inflammation, often resulting in delayed recovery and postponement of subsequent oncological treatment. In severe cases, these complications may be life-threatening.

Patients with a small main pancreatic duct (3 millimeters or less) are known to have a substantially higher risk of developing POPF. Previous studies have shown that several existing interventions may reduce the risk or severity of these complications. These include hydrocortisone, a medication that suppresses postoperative inflammation; octreotide, a medication that reduces the production of pancreatic secretions; and a surgical technique known as the ligamentum teres hepatis patch, which uses the patient's own tissue to protect nearby blood vessels in the event of a pancreatic leak.

Because the development of pancreatic fistulas is multifactorial, the investigators hypothesize that a combined approach targeting different underlying mechanisms may provide a complementary and more effective protective effect than any single intervention alone. The PANENCA trial therefore evaluates whether the combined use of hydrocortisone, octreotide, and the ligamentum teres patch can reduce the rate of major postoperative complications after pancreatoduodenectomy.

Patients participating in the study are randomly assigned to receive either the combination treatment in addition to standard perioperative care or standard perioperative care alone. The study medications are administered only during the first postoperative days, and the surgical patch is applied during the operation itself. No additional tests, monitoring procedures, or hospital visits are required beyond routine clinical care.

This international, multicenter randomized trial includes patients at high risk for POPF who are undergoing pancreatoduodenectomy. The primary objective is to determine whether the combination treatment reduces the incidence of major postoperative complications. If proven effective, this bundle approach may be implemented more consistently across participating countries and incorporated into international clinical guidelines for pancreatic surgery.

DETAILED DESCRIPTION:
The PANENCA trial is an international, multicenter, randomized controlled superiority trial designed to evaluate whether a standardized perioperative bundle approach reduces major postoperative complications in patients undergoing pancreatoduodenectomy who are at high risk for postoperative pancreatic fistula (POPF). High risk is defined preoperatively by a small main pancreatic duct diameter (≤3 mm) on cross-sectional imaging, which is associated with soft pancreatic parenchyma and an increased risk of anastomotic failure.

POPF remains the leading cause of morbidity and mortality following pancreatoduodenectomy. Several low-cost and widely available interventions have individually demonstrated effectiveness in reducing POPF or its sequelae; however, these measures have not been implemented consistently, systematically evaluated in a large international randomized trial, nor combined into a standardized perioperative strategy. The PANENCA trial therefore evaluates a bundled intervention (the HOP bundle) consisting of the following components:

1. Hydrocortisone, administered intravenously starting during induction of anesthesia to attenuate the postoperative inflammatory response, which is considered a key contributor to the development of POPF. Hydrocortisone is administered at a dose of 100 mg three times daily for three days, resulting in a total of 9 doses.
2. Octreotide, administered subcutaneously starting during induction of anesthesia, to reduce exocrine pancreatic secretion during the early postoperative period. Octreotide is administered at a dose of 0.1 mg three times daily for up to seven days or until earlier discharge, with a maximum of 21 doses.
3. A ligamentum teres hepatis patch, applied intraoperatively to mechanically protect the gastroduodenal artery stump from enzymatic erosion in the event of a POPF. The ligamentum teres is positioned between the gastroduodenal artery stump and the pancreatojejunostomy, functioning as an interpositional layer or wrap around one or both structures.

These interventions have potential complementary and non-overlapping mechanisms of action and are supported by prior randomized trials and meta-analyses. All investigational medicinal products are authorized and are used within approved or evidence-based indications.

Eligible patients are randomized in a 1:1 ratio prior to surgery to receive either the HOP bundle in addition to standard perioperative care or standard perioperative care alone. Randomization is stratified by participating center to account for potential inter-center variability. The trial is classified as a low-interventional clinical trial according to the European Union Clinical Trials Regulation (EU No 536/2014), as it uses authorized medicinal products, evidence-based dosing regimens, and does not require additional diagnostic or monitoring procedures beyond standard clinical practice.

Patients are followed from the day of surgery until hospital discharge, with additional follow-up to 90 days postoperatively for assessment of postoperative complications, readmissions, and mortality. No additional outpatient visits or diagnostic procedures are mandated beyond routine postoperative care.

The trial is powered to detect a superiority effect of the HOP bundle on the primary endpoint of major postoperative complications. Sample size calculations are based on contemporary national audit data demonstrating a substantially higher complication rate in patients with small pancreatic ducts. Allowances are made for intraoperative non-resection due to metastatic disease and for minimal loss to follow-up. A predefined interim analysis for futility and safety is planned. Detailed statistical methodology, including handling of missing data and definition of analysis populations, is specified in the statistical analysis section of the protocol.

Data are collected prospectively using a standardized electronic case report form (eCRF). Variables collected include baseline characteristics, intraoperative details, postoperative outcomes, and adverse events, all of which are routinely recorded as part of standard surgical care. Definitions of postoperative complications follow internationally accepted criteria, including those of the International Study Group of Pancreatic Surgery (ISGPS).

Data quality is ensured through predefined range and consistency checks within the eCRF system, central data monitoring, and on-site or remote monitoring in accordance with Good Clinical Practice (GCP). Source data verification is performed on a risk-based basis by comparison with medical records and operative reports. Serious adverse events and suspected unexpected serious adverse reactions are reported in accordance with regulatory requirements and overseen by an independent Data Safety Monitoring Board.

Both hydrocortisone and octreotide have well-established safety profiles. Given the short duration and low dosing used in this trial, the additional risk to participants is considered minimal. Postoperative monitoring, including glucose monitoring and routine laboratory assessments, follows standard clinical practice. Criteria for temporary trial suspension or early termination are predefined, and safety oversight is provided by an independent monitoring committee.

The study is conducted in accordance with the Declaration of Helsinki, International Council for Harmonisation Good Clinical Practice (ICH-GCP), and applicable national and European regulations. Written informed consent is obtained from all participants prior to enrollment. Patient representatives were involved in the design of the trial and will remain engaged throughout its conduct and dissemination of results.

Upon completion, study results will be submitted for publication in peer-reviewed journals and presented at international scientific meetings. A summary of results will be made publicly available in accordance with applicable transparency regulations.

ELIGIBILITY:
Inclusion Criteria:

* Elective pancreatoduodenectomy for any indication (both minimally invasive and open)
* Pancreatic duct diameter ≤ 3mm on preoperative CT or MRI*
* 18 years of age or older
* Signature of informed consent
* In the opinion of the investigator, the patient is eligible for the administration of hydrocortisone and octreotide, based on contraindications, warnings, and precautions as listed in the respective SmPCs

Exclusion Criteria:

* Age < 18 years
* Pregnancy or current breastfeeding
* Known allergy or hypersensitivity to hydrocortisone or octreotide
* Systemic fungal infection
* Concomitant use of strong CYP3A4 inhibitors or moderate-to-strong inducers that cannot be discontinued (see CYTOCHROME P450 DRUG INTERACTION TABLE (iu.edu))

  * Inhibitors must be discontinued ≥7 days before randomization
  * Inducers must be discontinued ≥28 days before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Major complications | Until postoperative day 90
  Rate of Major Complications, defined as a Clavien-Dindo score of ≥III and/or postoperative abdominal drain placement

SECONDARY OUTCOMES:
Postoperative Pancreatic Fistula (POPF) | Until postoperative day 90
  Rate of POPF grade B/C

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided